CLINICAL TRIAL: NCT06883760
Title: Intervention Study on Probiotic Composite Compressed Candy Tablets for Alleviation of Alcohol-Induced Symptoms
Brief Title: Intervention Study on Probiotic Combination Tableted Candy Hangover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Fengqin Feng, professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LL2023-X27
Record Dates: First submitted 2025-03-06; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Probiotic Combination Have the Potential to Improve Alcohol and Acetaldehyde in the Body After Drinking; The Potential of the Probiotics Combination Tablet on Alcohol Metabolism
Keywords: probiotics; medicine and food homologous substances; bioactive peptides; alcohol consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Probiotic tablet candy group
- Probiotic tablet candy (Experimental)
  Interventions: Combination Product: Probiotic tablet candy group

INTERVENTIONS:
Combination Product: Probiotic tablet candy group — 40 volunteers were randomly divided into two groups (n=20): Group A (probiotic → washout → placebo) and Group B (placebo → washout → probiotic). Each group took 1g of tablets (0.5g/tablet, 2 tablets) twice daily for 1 week, followed by a 2-week washout, then switched interventions. Fecal samples were collected at baseline, Day 7, and Day 28. Alcohol tests were conducted on Days 7 and 28 after fasting; participants consumed alcohol (1 mL/kg, 40% v/v) with a standard meal. Serum and saliva were collected post-meal. Body weight was measured, and alcohol dosage was adjusted accordingly. Participants maintained their usual diet and avoided alcohol-detoxifying or liver-protecting drugs. Medication during alcohol tests: 2 pills before tolerance test (after lunch), 2 pills before drinking, and 2 pills after waking.

SUMMARY:
Study Design Type: Randomized, blinded, placebo-controlled, crossover trial Participants: 40 volunteers, divided into two groups (n=20) Grouping Method: Minimization randomization based on age and BMI matching

Intervention Sequence:

Group A: Probiotic intervention → washout → placebo intervention Group B: Placebo intervention → washout → probiotic intervention Blinding: Participants, data collectors, and data analysts were blinded Roles: Randomization, data collection, and data analysis were performed by different researchers

Intervention Process

Phase 1 (Week 1):

Group A: Took probiotic tablets (1g twice daily, 0.5g/tablet) Group B: Took placebo tablets (1g twice daily, 0.5g/tablet) Washout Period: 2 weeks

Phase 2 (Week 4):

Group A: Took placebo tablets Group B: Took probiotic tablets

Sample Collection

Fecal Samples: Collected at three time points:

Baseline (1 week before alcohol test) Day 7 (after Phase 1) Day 28 (after Phase 2) Alcohol Tests: Conducted on Day 7 and Day 28 after overnight fasting Body Weight: Measured on test days; alcohol dosage adjusted accordingly (1 mL/kg, 40% v/v) Serum and Saliva: Collected at multiple time points post-alcohol consumption

DETAILED DESCRIPTION:
A randomized, blinded, placebo-controlled, crossover trial was conducted. Forty participants were divided into two groups (n=20). Then, for each block, randomization was performed by minimization by matching age and body mass index (BMI). The two groups received different sequences of Probiotic combination intervention and maltodextrin intervention (placebo), coded as A and B to conceal their identities. Participants, data collectors, and data analysts were blinded throughout the study. Different researchers performed randomization, data collection, and data analysis.

The 40 volunteers recruited were randomly divided into two groups (n=20) after signing the informed consent form, namely the Probiotic combination intervention group (Group A, probiotic intake → flushing → placebo intake) and the maltodextrin (placebo) group (Group B, placebo intake → flushing → probiotic intake). Group A tried the compressed tablet product for 1 week, and Group B tried the placebo for 1 week; after a 2-week washout period, Group A tried the placebo for 1 week, and Group B tried the compressed tablet product for 1 week. During the intervention period, volunteers took 1g of the compressed tablets twice a day (0.5g/tablet, 2 tablets) in the morning, noon and evening, and during the intervention period, volunteers took 1g of the placebo twice a day (0.5g/tablet, 2 tablets) in the morning and evening. Feces of all volunteers were collected one week before the alcohol experiment (first time), and the second and third feces were collected on the 7th and 28th days, respectively. Alcohol tests were performed on the 7th and 28th days after an overnight fast. Body weight was measured on the test day, and liquor was provided according to body weight. Participants ate a meal (standard diet) containing alcohol (alcohol content: 40% v/v, 1 mL/kg body weight), and serum and saliva of volunteers were collected at different time points after the meal. During the intervention period, all subjects followed their original dietary habits and stopped taking other alcohol-detoxifying and liver-protecting drugs or drugs that may affect alcohol metabolism. The medication method during the alcohol test was: 2 pills before the alcohol tolerance test after lunch (the first time point); 2 pills before drinking (i.e., before the hangover test at two time points); and 2 pills after waking up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years old
* BMI: 18-25 kg/m2
* Healthy adults with experience of being drunk, fully understanding the experimental plan, and voluntarily agreeing to participate
* Able to tolerate a certain amount of alcohol (calculated as 60 kg, about 60 mL of 40-proof liquor)
* Must be able to swallow tablets

Exclusion Criteria:

* People who are very intolerant to alcohol, with aldehyde dehydrogenase activity of 2%
* People with a history of allergic reactions or clinical allergic reactions to drugs, alcohol, products or other ingredients
* People who have taken drugs that induce and inhibit drug metabolizing enzymes, such as barbiturates, within one month from the date of the screening test
* People who have taken drugs that affect the results of clinical trials (alcohol metabolism) (aspirin, antipyretics, anti-inflammatory drugs, analgesics, antibiotics, herbal medicines, oral steroids, hormones, etc.) within 1 month from the screening population
* People who have taken drugs, products and functional foods that affect the intestines (such as probiotics, yogurt, etc.) within 10 days before the test
* People who have taken drugs, products or functional foods that have a functional effect on the stomach and liver within 10 days before the test
* People who have taken drugs, products or functional foods that have a functional effect on the stomach and liver within 10 days before the test. Those who have taken products that affect the test results, such as products or drugs that relieve alcohol, etc.
* Those who suffer from severe acute or chronic diseases such as cardiovascular disease, metabolic disease, hepatobiliary disease, pancreatic disease, muscle disease, nervous system disease, mental disorder, endocrine disease, immune disease, kidney disease, malignant tumor, lung disease and other diseases that require treatment
* Those who have received or are receiving clinically significant treatment for gastrointestinal diseases such as gastric or duodenal ulcers
* Those who have donated blood within 2 months from the date of screening
* Those whose serum AST, ALT or creatine kinase levels are higher than the reference range or twice the serum upper limit, and the creatinine level in the diagnostic test exceeds 2.0 mg/dL
* Those who are considered unsuitable due to diagnostic test results or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline blood alcohol during alcohol test at 1 month | Baseline (Day 0), Intervention end point (Day 28)
  Determination of the change of blood alcohol of the participants during alcohol test at 1 months.

SECONDARY OUTCOMES:
Changes in serum acetaldehyde during alcohol test at 1 month | Baseline (Day 0), Intervention end point (Day 28)
  Determination of the changes of serum acetaldehyde during alcohol test at 1 month
Changes of saliva acetaldehyde during alcohol test from baseline at 1 month | Baseline (Day 0), Intervention end point (Day 28)
  Determination of the changes of saliva acetaldehyde during alcohol test from baseline at 1 month
Change from baseline fecal microbiota at 1 month | Baseline (Day 0), Intervention end point (Day 28)
  Determination of the change from baseline fecal microbiota at 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- ZJUT(Zhejiang University of Technology), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Privacy and Ethical Concerns: IPD often contains sensitive personal information, and sharing it may violate privacy protection regulations or the requirements of ethical review boards, especially if the data is not fully de-identified.
  Data Ownership and Control: The research team may retain ownership of the data and wish to maintain control over its use to ensure it is utilized in alignment with the original research objectives.
  Intellectual Property and Commercial Interests: Certain research may involve potential commercial value or intellectual property, and sharing IPD could impact future patent applications or commercialization efforts.
  Resource Constraints: Preparing and sharing IPD in a usable and compliant format can be time-consuming and resource-intensive, which may not be feasible for the research team.
  Risk of Misinterpretation: Shared data might be misinterpreted or misused by others, potentially leading to incorrect conclusions or misuse of the findings.